CLINICAL TRIAL: NCT01802164
Title: Prophylactic Mesh Implantation in Patients With Peritonitis for the Prevention of Incisional Hernia: A Randomized Controlled Trial
Brief Title: Prophylactic Mesh Implantation in Patients With Peritonitis for the Prevention of Incisional Hernia
Acronym: PerProMe
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems due to very restricted inclusion criteria
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 006/12
Record Dates: First submitted 2013-02-15; First posted 2013-03-01 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Peritonitis; Incisional Hernia; Surgery
MeSH Terms: conditions — Peritonitis; Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Conventional abdominal wall closure with mesh implantation
  Interventions: Device: A non-absorbable composite mesh (Ethicon Physiomesh)
- 2 (No Intervention): Conventional abdominal wall closure without mesh implantation

INTERVENTIONS:
Device: A non-absorbable composite mesh (Ethicon Physiomesh) — To compare prophylactic mesh implantation to conventional abdominal wall closure in patients undergoing emergency laparotomy for peritonitis.
  Arms: 1

SUMMARY:
In patients undergoing laparotomy, the incidence of abdominal wall related complications such as incisional hernia is very high. In particular in patients with peritonitis undergoing laparotomy the incidence of incisional hernia is up to 54.3%. Furthermore, these patients are at great risk for development of postoperative fascial dehiscence.

The gold standard of abdominal wall closure is a running slowly absorbable suture irrespective of the presence of peritonitis. Implantation of an intraperitoneal mesh potentially reduces the incidence of incisional hernia.

In a series of high risk patients in which we implanted non-absorbable intraperitoneal mesh prophylactically we reduced the incidence of incisional hernia down to 3.2%.

DETAILED DESCRIPTION:
Background

Incisional hernia is a common complication in visceral surgery and varies between 11 and 26% in the general surgical population [1,2]. An incisional hernia is defined as any abdominal wall gap with or without a bulge in the area of postoperative scar perceptible or palpable by clinical examination or imaging [3]. Overall incidence of incisional hernia at our institution with a follow-up of five years was 14%, whereas in patients undergoing liver transplantation we found an incidence of incisional hernia of 25% in a prospective study [2]. However, patients with peritonitis are at very high risk for the development of incisional hernia. Moussavian et al demonstrated an incidence of incisional hernia of 54.3% after a median follow-up of 6 years in patients undergoing emergency surgery for secondary peritonitis [4]. In patients undergoing surgical therapy for secondary peritonitis, redo surgery because of complications associated with the abdominal wall, such as fascial dehiscence and surgical site infection are frequent. Impaired wound healing in response to the systemic inflammatory response and the high incidence of surgical site infection might render the abdominal wall even more susceptible for incisional hernia, compared with the general surgical population [5,6]. Furthermore, patients with peritonitis undergoing emergency laparotomy develop fascial dehiscence in up to 24.1% [7]. Fascial dehiscence requires reoperation and is associated with a mortality rate up to 44% [8].

Objective

To compare prophylactic mesh implantation to conventional abdominal wall closure in patients undergoing emergency laparotomy for peritonitis.

Methods

Implantation of a non-resorbable intraperitoneal mesh in patients with peritonitis undergoing emergency laparotomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical signs of peritonitis
* Emergency laparotomy or laparoscopy with conversion to laparotomy
* Patients > 18 years
* Written informed consent

Exclusion Criteria

* Previous implanted mesh
* Incisional hernia present
* Small bowel obstruction without bowel resection
* Surgery for cholecystitis
* Inflammatory bowel disease (Crohn's disease, Ulcerative colitis)
* Polytrauma patients
* Pregnant women
* Women younger than 45 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with incisional hernia | 54 months

SECONDARY OUTCOMES:
Number of patients with facial dehiscence | 54 months
Mortality | 54 months
Number of patients with surgical site infection | 54 months
Number of patients with intestinal fistula | 54 months
Number of patients with small bowel obstruction | 54 months
Number of patients with postoperative pain | 54 months
Number of patients with low grade mesh infection or chronic subclinical inflammation | 54 months
Number of patients with mesh explantation | 54 months

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, Prof. Dr. med., Principal Investigator — Dep. of visceral and transplant surgery; Univesrity Hiospital, Berne
Locations (1):
- Dep. of visceral and transplant surgery, Berne University Hospital, Bern, Canton of Bern, Switzerland